CLINICAL TRIAL: NCT00232414
Title: A Double-Blind Randomized Placebo Controlled Study of Quetiapine for the Treatment of Depression in Adolescents With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Melissa Delbello, Professor, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRUSQUET0384
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Bipolar I Disorder
Keywords: bipolar; with acute depressive episode
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
In this study, quetiapine is being tested for the possible treatment of bipolar I disorder with an acute depressive episode in children and adolescents.

We hypothesize that quetiapine will be more efficacious than placebo for the treatment of episodes of major depression associated with adolescent BP. Moreover, we hypothesize that quetiapine will be safe and well-tolerated compared with placebo for the treatment of depression associated with adolescent BP. Based on data from the BOLDER study and other studies of atypical antipsychotics in patients with bipolar depression (Calabrese et al., 2004, Macfadden et al., 2004, Tohen et al., 2004), which in general reveal effect sizes of approximately 0.5, a conservative sample size calculation, assuming power of .8, estimates we would need approximately 15 patients in each group to identify a statistically significant group difference in our main outcome measure, change form baseline to endpoint in the Children's Depression Rating Scale (Poznanski, 1979).

DETAILED DESCRIPTION:
This is a double-blind, randomized 56-day treatment trial of quetiapine vs. placebo for the treatment of bipolar adolescents with acute depression. Randomization will be stratified by sex, the presence of psychotic features, and a site specific randomization schedule will be determined. Stratification of randomization by sex is necessary to control for the higher rate of co-occurring ADHD in males than in females with bipolar disorder. Bipolar disorder with ADHD may be more treatment refractory than bipolar disorder without ADHD. Stratification by the presence of psychosis is necessary to avoid all patients with psychosis being assigned to one treatment group. A randomization schedule will be developed by the Children's Hospital Medical Center Investigational Pharmacy.

Procedures Thirty adolescents who are hospitalized for an episode of major depression associated with BP, type I, (ages 12-18) will be recruited for the study over two years.

After providing informed consent (the parent or legal guardian), informed assent (the child), and signing the document (both the parent and the child), subjects will be evaluated using the Washington University at St. Louis Kiddie-Schedule for Affective Disorders and Schizophrenia (K-SADS, Geller et al., 1998) by raters with extensive training in the instrument and established inter-rater reliability (ICC>0.9) (DelBello et al., 2004). The WASH-U K-SADS is a semi-structured clinical interview with established validity and reliability to assess the presence of DSM-IV Axis I psychiatric disorders in children and adolescents (Geller et al., 1998). The K-SADS involves an interview with the child and another interview with the parent.

If the diagnosis of bipolar disorder, type I, current episode depressed is confirmed by the K-SADS, the following scales will also be performed:

1. The Children's Depression Rating Scale (CDRS) to assess the severity of depressive symptoms (Poznanski et al., 1979);
2. The Young Mania Scale (YMRS) to assess the severity of manic symptoms (Fristad et al., 1992; Young et al., 1978);
3. The Hamilton Anxiety Rating Scale (HAM-A) to assess the severity of anxiety symptoms (Hamilton, 1959)
4. The Clinical Global Impression Scale BP Version (CGI-BP) to quantify the child's overall baseline functioning (National Institute of Mental health, 1985); The CGI-BP is used by the clinician to record the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). At all visits following baseline, we will also perform the CGI-BP Improvement Scale to quantify the change from baseline in overall functioning. The score ranges from 1 (very much improved) to 7 (very much worse).
5. The Simpson-Angus Scale (Simpson and Angus, 1970), Barnes Akathisia Scale (Barnes 1989) and Abnormal Involuntary Movement Scale (AIMS, US Department of Health, 1976) to assess for extrapyramidal symptoms.

Patients who received prior treatment with lithium or valproate must have serum concentrations of <0.4 mEq/L and 50 mg/L respectively before receiving quetiapine or placebo. Patients treated with antipsychotics (po or IM, non-depot), stimulants, or other mood stabilizers must have a 48 hr. interval without receiving these agents prior to randomization, except for patients recently (within one dosing interval) treated with depot antipsychotics, who will be excluded from this trial. Patients treated with prior antidepressants must have a 7 day washout period (patients treated with fluoxetine will be excluded from this trial because of its long half-life).

Medication in this study will be administered in a double-blind manner. Patients randomized to quetiapine will be administered beginning at day 0, a dose of 100mg/day which will be titrated to 300mg/day by day 3, with flexible titration to 600mg/day (in 100mg/day increments) until day 28.

Patients will be evaluated by a blinded (to treatment status and adverse events) rater at baseline (day 0) (MPD), prior to being randomized to placebo or quetiapine. Ratings 1-4 will be done at baseline (day 0) and on days 7, 14, 21, 28, 35, 42, 49, and 56 (or termination from the study).

Extrapyramidal rating scales and adverse events will be assessed on days of efficacy ratings by a different rater from the rater who is performing rating scales. Adverse events will be evaluated by open-ended questions about side effects and by vital sign measures. Adverse events will be monitored, documented and tabulated by occurrence, frequency and severity. Any extrapyramidal symptoms that develop in patients will be appropriately treated via dose reduction and/or administration of anticholinergic agents (e.g. benztropine), and this will be recorded. Patients will receive no other psychotropic agents during the study except for lorazepam, as needed for anxiety or agitation, up to 4 mg/d for days 0-6, 2 mg/d on days 7 to 14, and 1mg/day on days 14-21. The doses of lorazepam administered to patients will be recorded. Patients requiring other psychotropic medications will be terminated at the point at which such interventions are required. Please see Table 1 for schedule of assessments and laboratory tests.

Investigators will be responsible for monitoring the safety of patients who have entered this protocol and for alerting AstraZeneca to any event that seems unusual, even if this event may be considered an unanticipated benefit to the patient. Additionally, baseline medical history, physical examination, laboratory tests, and vital signs (blood pressure, pulse, weight, height and temperature) will be performed. Blood pressure and pulse will be taken after a patient has been lying down for 5 minutes (supine) and after standing for approximately 2 minutes (standing). Laboratory tests will include a urine pregnancy test and serum complete blood count (CBC), liver function tests (LFTs), thyroid stimulating hormone (TSH), renal profile, prolactin level, fasting glucose, fasting lipid profile, and an EKG. Vital signs, including Body Mass Index (BMI) and waist circumference will be repeated on days 7, 14, 21, 28, 35, 42, 49, and 56 (or endpoint). All other labs will be performed at baseline (day 0) and day 56 (or termination from the study), with the exception of fasting plasma glucose, fasting plasma lipid profile, and complete blood count, which will also be repeated at day 28 (and days 0 and 56). A funduscopic and physical exam will be performed prior to and at termination of trial.

If at any point during the study if a patient has a CDRS suicide item score > one point higher than their baseline for any one week, or a score of > 3 they will be withdrawn from the study. Additionally, patients will be withdrawn from the study (and treated as clinically indicated) if they have a worsening of symptoms at day 14 or later, as indicated by a CGI-I score of > 6 or more at any time during the study or a minimal worsening of symptoms at day 21 or later as indicated by a CGI-I score of > 5 at 2 consecutive visits, starting at day 14.

Additionally, if at any point during the study patients has a CBC with differential that shows an Absolute Neutrophil Count (ANC) < 1.0 x 10-9/L, we will repeat the test within 24 hours, if it remains < 1.0 x 10-9/L, the patient will be discontinued from the study.

Patients will be discharged form the hospital when they are felt to be clinically stable as determined by their inpatient attending and treatment team in collaboration with Dr. DelBello.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, subjects must meet the following criteria:

1. Male or female patients, 12-18 years of age.
2. Female patients of menarche must be using a medically accepted means of contraception (e.g. oral contraceptives, Depo-Provera, abstinence).
3. Each patient's authorized legal guardian must understand the nature of the study and must provide written informed consent. Each patient must also give assent to study participation.
4. Patients must have a diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) BP, type I and currently display an acute depressive episode as determined by K-SADS (Geller et al 2000).
5. Patients must have a baseline (day 0) CDRS score of at least 40.
6. Subjects should be fluent in English.

Exclusion Criteria:

Patients will be excluded from the protocol for any of the following reasons:

1. Female patients who are either pregnant or lactating.
2. Clinically significant or unstable hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, hematologic or other systemic medical conditions.
3. Any history of current or past diabetes that was treated with pharmacological intervention.
4. Neurological disorders including epilepsy, stroke, or severe head trauma.
5. Clinically significant laboratory abnormalities, on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, lipid profile, fasting glucose, urinalysis, thyroid indices and EKG.
6. Depression due to a general medical condition or substance-induced depression (DSM-IV).
7. Mental retardation (IQ <70).
8. YMRS score of > 12.
9. History of hypersensitivity to or intolerance of quetiapine.
10. Prior history of quetiapine non-response.
11. DSM-IV substance (except nicotine or caffeine) dependence within the past 3 months.
12. Judged clinically to be at suicidal risk (defined as having active suicidal ideation, intent or plan, or a serious suicide attempt within 30 days, or a baseline CDRS suicide score of > 3).
13. Participation in a clinical trial of another investigational drug within 1 month (30 days) prior to study entry.
14. Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections and day 0.
15. Treatment with concurrent mood stabilizers or anticonvulsants, benzodiazepines (except as described below), psychostimulants, guanethidine, or guanadrel, or antidepressants.
16. Patient who were treated with carbamazepine at any point during the month prior to screening.
17. Schizophrenia or other psychotic disorders (including schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder, psychotic disorder not otherwise specified) as defined in the DSM-IV.
18. Major depressive disorder, dysthymic disorder, depressive disorder not otherwise specified.
19. Subjects who are not fluent in English.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Children's Depression Rating Scale (CDRS): Measure of efficacy will be a change in CDRS total scores from baseline endpoint.

SECONDARY OUTCOMES:
Secondary Efficacy Measures
CDRS response rate: Defined by a > 50% decrease from baseline to endpoint in CDRS total score.
Clinical Global Impression Improvement Scale BP Version (CGI-I BP) Improvement Score response rate: Defined by an endpoint CGI-I score of 1 or 2 (much or very much improved)
Hamilton Anxiety Rating Scale (HAM-A): Measure of efficacy will be change from baseline to endpoint in HAM-A
Safety
Proportion of patients who met criteria for treatment-emergent mania (YMRS score > 16 on two consecutive visits or at final assessment).
Incidence of adverse events
Incidence of EPS (as measured by change from baseline to endpoint in EPS rating scales)
Change from baseline to endpoint in all laboratory measures and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DelBello, MD, Principal Investigator — University of Cincinnati and Cincinnati Children's Hospital
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Danielyan A, Patino LR, Benanzer T, Blom TJ, Welge JA, Chang KD, Adler CM, DelBello MP. Cognitive, Family, and Quality-of-Life Characteristics of Youth with Depression Associated with Bipolar Disorder. J Child Adolesc Psychopharmacol. 2023 Aug;33(6):225-231. doi: 10.1089/cap.2023.0002. PMID 37590017